CLINICAL TRIAL: NCT03105583
Title: A Cross-sectional Study Evaluating Pregnancy Related Use of Vitamins and Medication
Acronym: PREVIM
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Michael Ceulemans, Pharm D - PhD Researcher, KU Leuven
Other Study IDs: MC201602
Record Dates: First submitted 2016-11-08; First posted 2017-04-10 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Medication and Supplement Use; Pregnant Women
Keywords: Medication beliefs; Information desire; Vitamin deficiencies
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women visiting the obstetrics department
  Interventions: Drug: Medication use during pregnancy; Dietary Supplement: Supplement use during pregnancy; Other: Vitamin status of a pregnant woman

INTERVENTIONS:
Drug: Medication use during pregnancy
Dietary Supplement: Supplement use during pregnancy
Other: Vitamin status of a pregnant woman — Haemoglobin, RBC count + hematocrits, thrombocytes count, folate (serum), vitamin B12, WBC count, ferritin, iron (serum), transferrin % and saturation, TSH, T4, free glucose, LDH, ALT, AST, GGT, bilirubin (total), CRP, albumin, total protein, ureum, uric acid, creating, calcium (total), 25-hydroxy vitamin D, Na, K, Mg

SUMMARY:
This cross-sectional study will try to give answers to the following project aims:

* To provide an overview of the prevalence of health products' use among Belgian pregnant women (prescription and OTC medication, vitamin supplements, phyto-therapeutics, dermatologic products), including where pregnant women buy or get their health products (online web survey).
* To document women's beliefs about medication during pregnancy and their information desire (online web survey).
* To determine the current vitamin status among pregnant women and to reveal clinical targets for supplementing deficiencies in this population (blood sample analysis).

The study will be performed at the obstetrics department of the University Hospitals of Leuven (campus Gasthuisberg).

We aim to include 300 pregnant women (100 per trimester), of which 150 women will be asked to determine their vitamin status (50 per trimester).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who visit the obstetrics department of the University Hospitals of Leuven
* ≥18 years
* Able to understand Dutch, French or English

Exclusion Criteria:

* <18 years
* Don't able to understand Dutch, French or English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who visit the obstetrics department of the University Hospitals of Leuven (campus Gasthuisberg) will be invited to participate, independent of their pregnancy trimester.
  Women can only participate once during their pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Medication and supplement use among Belgian pregnant women | Completion of a questionnaire during pregnancy: between 8-12weeks or 24-32weeks gestational age
  Percentage of women who have taken a health product during the last 7 days - Overview of the health products used by pregnant women

SECONDARY OUTCOMES:
Vitamin deficiencies among Belgian pregnant women | One blood sample during pregnancy: between 8-12weeks or 24-32weeks gestational age
  Analysis of a blood sample
Medication beliefs among Belgian pregnant women | Completion of a questionnaire during pregnancy: between 8-12weeks or 24-32weeks gestational age
  Beliefs about Medicines Questionnaire (BMQ) (R. Horne, H. Nordeng)

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Foulon, PhD, PharmD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No